CLINICAL TRIAL: NCT00228046
Title: Double-Blind, Placebo-Controlled Trial of Flexible Dose Divalproex Sodium Adjunctive to Stimulant Treatment for Aggressive Children With Attention-Deficit Hyperactivity Disorder
Brief Title: Medication Strategies for Treating Aggressive Behavior in Youth With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Joseph Blader, Stony Brook University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K23MH064975 (NIH); K23MH064975 (NIH); M01RR010710 (NIH); DSIR CT-M1
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2013-10-31 (Estimated); Status verified 2013-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Conduct Disorder; Oppositional Defiant Disorder
Keywords: ADHD; ODD; Conduct Disorder; CD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Conduct Disorder; Oppositional Defiant Disorder | interventions — Valproic Acid; Methylphenidate; Dextroamphetamine; Family Therapy

INTERVENTIONS:
Drug: Divalproex Sodium
Drug: Methylphenidate
Drug: Dextroamphetamine
Drug: Mixed Amphetamine Salts
Behavioral: Family Counseling
Behavioral: Behavior Management Training with Parents

SUMMARY:
This study will assess whether adding a mood stabilizer, divalproex sodium, to stimulant treatment is more effective than stimulant treatment alone in reducing aggressive behavior among children with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
ADHD is one of the most common childhood mental disorders. It often causes impaired functioning in multiple areas, including home, school, and peer relationships. Additionally, children with ADHD often develop aggressive behavior, which is not usually adequately suppressed by standard stimulant treatments for ADHD. In order to address this problem, many physicians prescribe multiple medications at once. There is no clinical evidence, however, proving that this method is safe and effective. This study will assess whether adding a mood stabilizer, divalproex sodium, to stimulant treatment is more effective than stimulant treatment alone in reducing aggressive behavior among children with ADHD.

Participants in this double blind study will first receive open label stimulant treatment for ADHD and a comorbid disruptive behavior disorder. Participants whose aggressive behavior subsides with stimulant treatment alone will not proceed into the next phase of the study. Participants whose ADHD symptoms lessen from the treatment but whose aggressive behavior persists will be randomly assigned to receive either divalproex sodium or placebo in addition to their stimulant treatment for 8 weeks. Study visits will be held weekly for 11 to 16 weeks. At these visits, aggression levels and medication side effects will be assessed. Families will also meet with the researchers to discuss the child's progress, and attend behavioral counseling with a therapist. Participants who did not continue into the second phase of the study will be asked to return to the study site for a follow-up visit 8 weeks following the end of the first phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ADHD
* Diagnosis of opposition defiant disorder or conduct disorder
* Score that exceeds the study threshhold on the standardized scale of aggressive behavior

Exclusion Criteria:

* Current psychosis
* Current major depression
* Current pervasive developmental disorder
* Current obsessive compulsive disorder
* Any other anxiety disorder as primary diagnosis
* Mental retardation

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2004-01; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Aggression (Measured by the Overt Aggression Scale after 8 weeks of treatment)
Improvement of ADHD symptoms (Measured by the Clinical Global Improvement Scale and ADHD Rating Scale after 8 weeks of treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph C. Blader, PhD, MSc, Principal Investigator — Stony Brook State University of New York School of Medicine
Locations (2):
- United States (2):
  - Long Island Jewish Medical Center / Schneider Children's Hospital, New Hyde Park, New York
  - Stony Brook University Hospital, Stony Brook, New York

REFERENCES:
- [Derived] Blader JC, Pliszka SR, Kafantaris V, Sauder C, Posner J, Foley CA, Carlson GA, Crowell JA, Margulies DM. Prevalence and Treatment Outcomes of Persistent Negative Mood Among Children with Attention-Deficit/Hyperactivity Disorder and Aggressive Behavior. J Child Adolesc Psychopharmacol. 2016 Mar;26(2):164-73. doi: 10.1089/cap.2015.0112. Epub 2016 Jan 8. PMID 26745211
- [Derived] Blader JC, Pliszka SR, Kafantaris V, Foley CA, Crowell JA, Carlson GA, Sauder CL, Margulies DM, Sinha C, Sverd J, Matthews TL, Bailey BY, Daviss WB. Callous-unemotional traits, proactive aggression, and treatment outcomes of aggressive children with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2013 Dec;52(12):1281-93. doi: 10.1016/j.jaac.2013.08.024. Epub 2013 Sep 25. PMID 24290461
- [Derived] Blader JC, Schooler NR, Jensen PS, Pliszka SR, Kafantaris V. Adjunctive divalproex versus placebo for children with ADHD and aggression refractory to stimulant monotherapy. Am J Psychiatry. 2009 Dec;166(12):1392-401. doi: 10.1176/appi.ajp.2009.09020233. Epub 2009 Nov 2. PMID 19884222